CLINICAL TRIAL: NCT06255600
Title: High-Definition Transcranial Direct Current Stimulation (Hd-Tdcs) and Chlorella Pyrenoidosa as an Adjuvant Treatment to Reduce Cardiovascular Risk in Patients With Long COVID
Brief Title: High-definition Transcranial Direct Current Stimulation and Chlorella Pyrenoidosa to Reduce Cardiovascular Risk
Acronym: HD-TDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: City University of New York (Other)
Responsible Party: Principal Investigator, Suellen Andrade, Suellen Marinho Andrade, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD-tDCS/Chlorella
Record Dates: First submitted 2024-02-11; First posted 2024-02-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases; Long Covid19
MeSH Terms: conditions — Cardiovascular Diseases; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Experimental group: Experimental group: Patients allocated to this group will receive a current of 3mA for 20 minutes of anodal HD-tDCS (4x1) for 10 sessions (twice a week in five weeks) and/or Chlorella Pyrenoidosa (5g/day), receiving 10 tablets per day for five weeks.
  Placebo/Sham Group: Patients allocated to this group will receive a simulated 3mA current with 30 seconds of acceleration and 30 seconds of deceleration minutes of anodal HD-tDCS (4x1) for 10 sessions (twice a week in five weeks) and/or Placebo with maltodextrin (5g/day) being 10 capsules per day for five weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research includes the responsible researcher, assistant and collaborator. Collaborating Researcher is responsible for applying the technique to the patient, knowing which stimulus will be true or placebo. He must apply the research tools and fill out the forms. Alert the main researcher and assistant regarding signs and symptoms in patients resulting from adverse effects.
  In this way, the patient and the collaborating researcher are blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental HD-tDCs (Experimental): Patients will be randomly enrolled into this group. They will receive stimulation in the portion of the left primary motor cortex (M1) by HD-tDCS (lasting 20 minutes of 4x1 tDCS-HD) with anodal stimulus, twice a week for five weeks. The electric current will be supplied with an acceleration time of 30 seconds and will be maintained for 20 minutes and then reduced by 30 seconds
  Interventions: Other: High Definition-transcranial Direct Current Stimulation
- Experimental HD-tDCS and Chlorella (Experimental): Patients will be randomly enrolled into this group. They will receive stimulation in the portion of the left primary motor cortex (M1) by HD-tDCS (lasting 20 minutes of 4x1 tDCS-HD) with anodal stimulus, twice a week for five weeks. The electric current will be supplied with an acceleration time of 30 seconds and will be maintained for 20 minutes and then reduced by 30 seconds. In addition, they will receive functional food that will be provided in the form of 10 tablets per day of Chlorella Pyrenoidosa (5g/day) containing 4mcg of B12, organically pressed into tablets (Registration with ANVISA/MS: 6.7273.000) for five weeks.
  Interventions: Other: High Definition-transcranial Direct Current Stimulation; Dietary Supplement: Chlorella Pyrenoidosa
- Experimental Chlorella (Experimental): Patients will be randomly enrolled into this group. They will receive the functional food that will be provided in the form of 10 tablets per day of Chlorella Pyrenoidosa (5g/day) containing 4mcg of B12, organically pressed into tablets (Registration with ANVISA/MS: 6.7273.000) for five weeks.
  Interventions: Dietary Supplement: Chlorella Pyrenoidosa
- Placebo/Sham (Sham Comparator): Patients allocated to this group will receive a simulated 3mA current with 30 seconds of acceleration and 30 seconds of deceleration minutes of anodal HD-tDCS (4x1) for 10 sessions (twice a week in five weeks) and/or Placebo with maltodextrin (5g/day) being 10 capsules per day for five weeks.
  Interventions: Other: High Definition-transcranial Direct Current Stimulation; Dietary Supplement: Chlorella Pyrenoidosa

INTERVENTIONS:
Other: High Definition-transcranial Direct Current Stimulation — High-Definition transcranial Direct Current Stimulation (HD-tDCS) is a neuromodulation technique, is non-invasive, targeted, safety.
  Arms: Experimental HD-tDCS and Chlorella; Experimental HD-tDCs; Placebo/Sham
Dietary Supplement: Chlorella Pyrenoidosa — functional food, organically pressed into tablets (Registration with ANVISA/MS: 6.7273.000)
  Arms: Experimental Chlorella; Experimental HD-tDCS and Chlorella; Placebo/Sham

SUMMARY:
Recent investigations have shown that of the patients who were affected by SARCov2 have remained with persistent symptoms in a high proportion. In these considerations, the literature has suggested nomenclatures such as "post-COVID-19" and "chronic COVID-19", "long -COVID" and Post-Covid Syndrome for patients recovered from SARCov2 reporting persistent symptoms and signs for weeks to months after resolution of the acute infection. Furthermore, there may be cardiovascular complications in affected patients, the consequences of which can lead to muscle contractility disorders, vascular insufficiency, cardiac arrest, reinforcing the need for controlled, randomized studies, as well as follow-up and monitoring of these. Furthermore, cardiovascular diseases (CVD) are part of the health problems that lead to the most deaths in the world, they also lead to a high proportion of hospital admissions, due to the worsening of the pathology and a higher incidence in the elderly population. The worsening of CVD conditions leads to inadequate food consumption at the hospital level, causing changes in several nutrients, including vitamin B12. The reduction in B12 levels leads to changes in several systems, including the cardiovascular system, and due to the increase in homocysteine and the triggering of the inflammatory cascade. Studies indicate that B12 supplementation through Chlorella (microalgae - functional food) reduced cardiovascular risk and modulated the inflammatory cascade. In combination, neurostimulation has presented aspects that promote pain neuromodulation, due to the improvement of respiratory patterns and inflammatory modulation. More specifically, there is a protocol with promoting findings, this being HD-tDCS. In this sense, this research aims to evaluate the effects of HD-tDCS and the consumption of Chlorella Pyrenoidosa to improve B12 levels in patients with cardiovascular risk post-COVID-19.

DETAILED DESCRIPTION:
This study is an open label research, clinical trial, double blind, placebo controlled, and randomized, involving assistance to patients at risk of cardiovascular disease, in outpatient care (Continue Caring Project). Included in the research are adults and elderly participants at cardiovascular risk, whose initial diagnosis for hospitalization was due to COVID-19 and at the hospital level those admitted for treatment in the Intensive Care Unit or ward with heart disease who are eligible for neurostimulation by HD-tDCS. Patients will be randomly allocated into an experimental and control group for HD-tDCS and also to receive the functional food. The protocol will be HD-tDCS (lasting 20 minutes of 4x1 tDCS-HD) positioning the central electrode in the left primary motor cortex (M1) with anodal stimulus, twice a week; nutritional monitoring; collection of laboratory tests (at the beginning and end of treatment) and the group that will receive the functional food will be provided with 10 tablets of Chlorella Pyrenoidosa (5g/day) containing 4mcg of B12, organic pressed into tablets (Registration with ANVISA/MS : 6,7273,000) for five weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiovascular diagnosis or risk;
* Adults and elderly people (18 to 80 years old);
* Able to respond to commands and grant consent to participate in the research through the informed consent form;
* Who have post-COVID symptoms.

Exclusion Criteria:

* Patients with a clinical history of neuromuscular or cognitive instability, pregnancy and contraindications for receiving neurostimulation (such as cardiac pacemakers and metallic brain implants);
* Patients with contraindications to the use of Chlorella (gastritis, esophagitis, peptic ulcers),
* Pregnant patients, patients with stroke and tumors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults and older adults
Enrollment: 60 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Change B12 by blood analysis biochemical | After five week of the group of research start
  Change B12 (above 148pmol/L)

SECONDARY OUTCOMES:
Change Methylmalonic Acid and Homocysteine | After five week of the group of research start
  Change blood levels of Methylmalonic Acid and Homocysteine (below 270nmol/L and 12mmol/L, respectively)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanessa Meira Cintra, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No